CLINICAL TRIAL: NCT03434977
Title: A Randomized, Open-Label, Cross-over Phase 1 Study to Evaluate the Food Effect of Single Oral Dose of TAK-536 Pediatric Formulation in Healthy Adult Male Subjects
Brief Title: A Phase 1 Food Effect Study of Azilsartan (TAK-536) Pediatric Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Azilsartan-1005; U1111-1206-5973 (Other: WHO); JapicCTI-183856 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-536 10 mg (fasted) + TAK-536 10 mg (fed) (Experimental): TAK-536 10 milligram (mg) granule formulation (pediatric formulation), once daily on Day 1 of Period 1 (6 days) in the morning under fasted condition, followed by wash-out (6 days), followed by TAK-536 10 mg granule formulation (pediatric formulation), once daily on Day 1 of Period 2 (6 days) after starting breakfast.
  Interventions: Drug: TAK-536
- TAK-536 10 mg (fed) + TAK-536 10 mg (fasted) (Experimental): TAK-536 10 mg granule formulation (pediatric formulation), once daily on Day 1 of Period 1 (6 days) after starting breakfast, followed by wash-out (6 days), followed by TAK-536 10 mg granule formulation (pediatric formulation), once daily on Day 1 of Period 2 (6 days) in the morning under fasted condition.
  Interventions: Drug: TAK-536

INTERVENTIONS:
Drug: TAK-536 — TAK-536 granule formulation

SUMMARY:
The purpose of this study is to assess the PK of TAK-536 and effect of food on the PK following single oral administration of TAK-536 pediatric formulation in Japanese healthy adult male participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-536. TAK-536 is being tested in Japanese healthy adult male participants. This study will look at the PK and effect of food on the PK following single oral administration of TAK-536 pediatric formulation.

The study will enroll 12 healthy participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups and will receive a single oral dose of 10 mg of TAK-536 pediatric formulation with 200 mL of water according to the following treatments in each period during the study.

* Treatment Group A: single oral administration in the morning under fasted condition (Period 1), followed by single oral administration after breakfast (Period 2)
* Treatment Group B: single oral administration after breakfast (Period 1), followed by in the morning under fasted condition (Period 2)

This single-center trial will be conducted in Japan. The overall time to participate in this study is approximately one month. Participants will make five visits to the clinic and be hospitalized for eight days in total.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a Japanese healthy adult male.
4. The participant ages 20 to 35 years inclusive at the time of informed consent.
5. The participant weighs at least 50.0 kilogram (kg), and has a Body Mass Index (BMI) between 18.5 and 25.0 kilogram per square meter (kg/m^2), inclusive, at Screening.

Exclusion Criteria:

1. The participant has suspected hypotension with associated physical findings, such as dizziness postural, facial pallor, or cold sweats based on evaluation/physical examination at Screening, on the day before the study drug administration (Day -1) in Period 1, or up to the study drug administration in Period 1.
2. The participant has received any study drug within 16 weeks (112 days) prior to the study drug administration in Period 1.
3. The participant has received TAK-536 or TAK-491 in a previous clinical study or as a therapeutic agent.
4. The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
5. The participant has a hypersensitivity to any component of the formulation of TAK-536 or any ARB.
6. The participant has a positive urine drug result for drugs of abuse (defined as any illicit drug use) at Screening.
7. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. The participant has taken any excluded medication, supplements, dietary products or food products during the specified time periods.
9. The participant has any current or recent (within 6 months prior to the start of the study drug administration in Period 1) gastrointestinal diseases that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention).
10. The participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1 of Period 1.
11. The participant has a positive test result for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at Screening.
12. The participant has poor peripheral venous access.
13. The participant has undergone whole blood collection of at least 200 milliliter (mL) within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of the study drug administration in Period 1.
14. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of the study drug administration in Period 1.
15. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of the study drug administration in Period 1.
16. The participant has an abnormal (clinically significant) ECG at Screening or prior to the study drug administration in Period 1.
17. The participant has abnormal laboratory values that suggest a clinically significant underlying disease, or participant with the following laboratory abnormalities at Screening or prior to the study drug administration in Period 1: Alanine Aminotransferase (ALT) and/or Aspartate Transaminase (AST) greater than (>) 1.5× the upper limits of normal (ULN).
18. The participant who, in the opinion of the investigator or sub-investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2018-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 14 February 2018 to 11 March 2018.
Pre-assignment Details: Healthy male participants were enrolled in 1 of the 2 treatment sequences of this 2-period cross-over study to receive pediatric formulation of TAK-536 10 milligram (mg) granules under fasted or fed condition.
Groups:
- TAK-536 10 mg Granules Fasted + TAK-536 10 mg Granules Fed: TAK-536 10 mg, granules (pediatric formulation), orally, under fasted condition, once on Day 1 of Period 1, followed by a washout period of at least 6 days, further followed by TAK-536 10 mg, granules (pediatric formulation), orally, under fed condition, once on Day 1 of Period 2.
- TAK-536 10 mg Granules Fed + TAK-536 10 mg Granules Fasted: TAK-536 10 mg, granules (pediatric formulation), orally, under fed condition, once on Day 1 of Period 1, followed by a washout period of at least 6 days, further followed by TAK-536 10 mg, granules (pediatric formulation), orally, under fasted condition, once on Day 1 of Period 2.
Period: Intervention Period 1 (6 Days)
Arm/Group | TAK-536 10 mg Granules Fasted + TAK-536 10 mg Granules Fed | TAK-536 10 mg Granules Fed + TAK-536 10 mg Granules Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (at Least 6 Days)
Arm/Group | TAK-536 10 mg Granules Fasted + TAK-536 10 mg Granules Fed | TAK-536 10 mg Granules Fed + TAK-536 10 mg Granules Fasted
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Intervention Period 2 (6 Days)
Arm/Group | TAK-536 10 mg Granules Fasted + TAK-536 10 mg Granules Fed | TAK-536 10 mg Granules Fed + TAK-536 10 mg Granules Fasted
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-536 10 mg Granules Fasted + TAK-536 10 mg Granules Fed | TAK-536 10 mg Granules Fed + TAK-536 10 mg Granules Fasted | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.7 (2.73) | 24.3 (5.57) | 23.5 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 6 | 6 | 12
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 175.7 (7.31) | 173.2 (5.71) | 174.4 (6.39)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 66.88 (5.712) | 64.02 (11.129) | 65.45 (8.566)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.72 (2.036) | 21.23 (2.392) | 21.47 (2.133)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 4 | 1 | 5
  Current smoker | 1 | 5 | 6
  Former smoker | 1 | 0 | 1
Alcohol Classification [Count of Participants; unit: Participants]
  Drank a few times per month | 5 | 5 | 10
  Never drank | 1 | 1 | 2
Caffeine Classification [Count of Participants; unit: Participants]
  Had caffeine consumption | 3 | 0 | 3
  Had no caffeine consumption | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The pharmacokinetic (PK) analysis set was defined as all participants who received the study drug, completed the minimum protocol-specified procedures without any major protocol deviations, and were evaluable for PK.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- TAK-536 10 mg Granules Fasted: TAK-536 10 mg, granules (pediatric formulation), orally, under fasted condition, once on Day 1 of either Period 1 or 2.
- TAK-536 10 mg Granules Fed: TAK-536 10 mg, granules (pediatric formulation), orally, under fed condition, once on Day 1 of either Period 1 or 2.
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
nanogram per milliliter (ng/mL) | 652.6 (78.03) | 609.4 (103.92)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were ratio of fed conditions divided by fasted conditions, taking anti-logs of the least square (LS) means difference (fed-fasted) or confidence interval (CI). The difference in LS means between treatment conditions (fed-fasted) and two-sided 90% CI were provided using a crossover analysis of variance (ANOVA) model. ANOVA model included log-transformed (natural log) PK parameters Cmax as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 0.937, 90% CI 2-sided [0.890 to 0.986]

2. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: The PK analysis set was defined as all participants who received the study drug, completed the minimum protocol-specified procedures without any major protocol deviations, and were evaluable for PK.
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
hours | 2.000 [1.00 to 4.00] | 3.000 [2.00 to 4.00]
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (non-natural log) PK parameters tmax as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; LS-Means Difference = 0.9083, 90% CI 2-sided [0.1821 to 1.6345]

3. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
hour*nanogram per milliliter (h*ng/mL) | 5275.3 (1044.49) | 5220.7 (881.13)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters AUClast as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 0.998, 90% CI 2-sided [0.943 to 1.056]

4. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
h*ng/mL | 5440.1 (1109.74) | 5377.8 (918.96)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters AUC∞ as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 0.997, 90% CI 2-sided [0.942 to 1.056]

5. Primary Outcome: T1/2z: Terminal Disposition Phase Half-life for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
hours | 11.11 (0.90050) | 10.96 (0.85065)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters T1/2z as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 0.985, 90% CI 2-sided [0.932 to 1.041]

6. Primary Outcome: MRTlast, ev: Mean Residence Time From Time 0 to the Time of the Last Quantifiable Concentration for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
hours | 9.419 (1.0233) | 9.836 (0.61518)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters MRTlast, ev as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 1.047, 90% CI 2-sided [1.006 to 1.091]

7. Primary Outcome: MRT∞, ev: Mean Residence Time From Time 0 to Infinity for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
hours | 11.02 (1.3931) | 11.40 (0.90089)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters MRT∞, ev as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 1.037, 90% CI 2-sided [0.996 to 1.081]

8. Primary Outcome: λz: Terminal Disposition Phase Rate Constant for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1 per hour (1/h)
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
1 per hour (1/h) | 0.06285 (0.0048845) | 0.06355 (0.0047738)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters λz as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 1.014, 90% CI 2-sided [0.959 to 1.071]

9. Primary Outcome: CL/F: Apparent Clearance for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter per hour (L/h)
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
Liter per hour (L/h) | 1.912 (0.40241) | 1.909 (0.31980)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters CL/F as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 1.003, 90% CI 2-sided [0.947 to 1.062]

10. Primary Outcome: Vz/F: Apparent Volume of Distribution for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 11
liter | 30.35 (5.5177) | 30.14 (5.2637)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules Fasted vs TAK-536 10 mg Granules Fed; The shown data were the ratio of the fed conditions divided by the fasted conditions, taking anti-logs of the LS means difference (fed-fasted) or CI. The difference in the LS means between treatment conditions (fed-fasted) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters Vz/F as dependent variable, and treatment condition, group, and period as independent variables; Test type: Other; Ratio = 0.989, 90% CI 2-sided [0.916 to 1.068]

11. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Baseline up to Day 18 (End of Period 2)
Population: The safety analysis set was defined as all participants who received at least one dose of the study drug. Out of 12 participants, only 11 participants received study drug under fasted condition, since 1 participant discontinued the study due to adverse event (AE) before the start of Period 2.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 12
Participants | 0 | 1

12. Secondary Outcome: Number of Participants With TEAE Related to Vital Sign
Time Frame: Baseline up to Day 18 (End of Period 2)
Population: The safety analysis set was defined as all participants who received at least one dose of the study drug. Out of 12 participants, only 11 participants received study drug under fasted condition, since 1 participant discontinued the study due to AE before the start of Period 2.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With TEAE Related to Body Weight
Time Frame: Baseline up to Day 18 (End of Period 2)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With TEAE Related to Clinical Laboratory Tests (Eosinophil Count Increased)
Time Frame: Baseline up to Day 18 (End of Period 2)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 12
Participants | 0 | 1

15. Secondary Outcome: Number of Participants With TEAE Related to 12-lead Electrocardiograms (ECGs)
Time Frame: Baseline up to Day 18 (End of Period 2)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
Number analyzed (Participants) | 11 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug until the follow up examination on Day 6 in Period 2 (Day 18)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
  Out of 12 participants, only 11 participants received study drug under fasted condition, since 1 participant discontinued the study due to AE before the start of Period 2.
Arm/Group | TAK-536 10 mg Granules Fasted | TAK-536 10 mg Granules Fed
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-536 10 mg Granules Fasted (N=11) | TAK-536 10 mg Granules Fed (N=12)
Eosinophil count increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03434977/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03434977/SAP_001.pdf